CLINICAL TRIAL: NCT05641870
Title: Molecular Profiling and Dynamic Changes of Circulating Tumor DNA in Unresectable Locally Advanced Non-small Cell Lung Cancer
Brief Title: Molecular Profiling and Dynamic Changes of ctDNA in Unresectable Locally Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Principal Investigator, Edurne Arriola, Principal Investigator, Parc de Salut Mar
Other Study IDs: 2022/10344/I
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer; Stage III Lung Cancer; Unresectable Lung Carcinoma
Keywords: Liquid biopsy; ctDNA; Chemoradiotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; Maintenance; Genome; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Biospecimen Retention: Samples With DNA — Tumor samples from tissue biopsy or citology. Whole blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sample collection — Tumor samples will be collected as standard diagnostic procedure at diagnosis. Plasma samples from whole blood extractions will also be collected at diagnosis, after chemoradiotherapy, and every 3 months from there until completing one year of follow-up.
Diagnostic Test: Characterization of the tumoral tissue genomic alterations — Genomic alterations of tumor tissue samples will be analyzed locally by next-generation sequencing when material is adequate, as standard diagnostic procedure.
Drug: Chemoradiation treatment regimen and maintenance (if amenable) — Patients will be treated with standard chemotherapy (following the clinical practice at each institution). Radiotherapy will be delivered concurrently when feasible with a total dose of 60-66 Gy. In selected cases, due to frailty of the patient or impaired pulmonary function, radiotherapy will be delivered sequentially. In tumors with positive PD-L1 expression, a year of durvalumab 10 mg/m2 every 2 weeks will be administered if there are no contraindications.
Diagnostic Test: Genomic and methylation analysis in liquid biopsy — Blood samples for ctDNA genomic and methylation analysis (4 mL of plasma for each sample) will be sent to the Guardant Health Laboratories in the US and analyzed after Contractual Agreement signature, using the Guardant Reveal test.
  This liquid biopsy test uses ctDNA to detect presence of MRD and monitor for recurrence after definitive surgical/systemic therapy for patients with cancer. It has been validated in early-stage colorectal cancer and integrates assessment of somatic alterations with an epigenomic cancer signature to identify the presence of methylation signatures associated with cancer versus normal DNA.

SUMMARY:
Multi-center observational clinical study to evaluate the application value of ctDNA monitoring in efficacy assessment and relapse prediction in patients diagnosed with unresectable, locally advanced NSCLC receiving CRT with or without durvalumab maintenance treatment.

DETAILED DESCRIPTION:
Newly diagnosed, histologically confirmed, unresectable stage III NSCLC patients, amenable to receive standard of care chemoradiotherapy with or without durvalumab maintenance, will be enrolled in this study. Whole blood collection will be conducted during the treatment for ctDNA detection in specific time-points of interest. Next-generation sequencing using commercially available panels, and analysis of ctDNA aberrant methylation will be performed. Results will be correlated to patients' recurrence times and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, histologically confirmed, unresectable locally advanced NSCLC.
* ≥18 years of age.
* Ability to understand the written informed consent and willingness to sign it.

Exclusion Criteria:

* Patients who are unwilling to follow-up evaluation of response to therapy.
* Any condition that, in the opinion of the investigator, would interfere with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, histologically confirmed, unresectable stage III NSCLC patients, amenable to receive standard of care chemoradiotherapy with or without durvalumab maintenance.
  Patients will be recruited in two centers: Hospital del Mar (Barcelona, Spain) and Instituto Português de Oncologia (Porto, Portugal). The expected number of enrolments is 30-40 patients per year per institution. All patients will be informed of the research nature of the study and will be included after written informed consent is provided.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative variation of aberrant methylated ctDNA concentrations before chemoradiotherapy, after chemoradiotherapy, and every 3 months during 1 year of follow-up. | 16 months
Correlation between patients' recurrence or progression, and quantitative detection of circulating tumour DNA (ctDNA) concentration. | 2 years
Concordance of ctDNA genomic alterations detected in peripheral blood samples, with those in matched tumour samples. | At diagnosis
Correlation between survival outcomes (progression free survival, overall survival) and quantitative detection of ctDNA genomic alterations or methylation status. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Arriola, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar - Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Ettinger DS, Wood DE, Aisner DL, Akerley W, Bauman JR, Bharat A, Bruno DS, Chang JY, Chirieac LR, D'Amico TA, Dilling TJ, Dowell J, Gettinger S, Gubens MA, Hegde A, Hennon M, Lackner RP, Lanuti M, Leal TA, Lin J, Loo BW Jr, Lovly CM, Martins RG, Massarelli E, Morgensztern D, Ng T, Otterson GA, Patel SP, Riely GJ, Schild SE, Shapiro TA, Singh AP, Stevenson J, Tam A, Yanagawa J, Yang SC, Gregory KM, Hughes M. NCCN Guidelines Insights: Non-Small Cell Lung Cancer, Version 2.2021. J Natl Compr Canc Netw. 2021 Mar 2;19(3):254-266. doi: 10.6004/jnccn.2021.0013. PMID 33668021
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Lindeman NI, Cagle PT, Aisner DL, Arcila ME, Beasley MB, Bernicker EH, Colasacco C, Dacic S, Hirsch FR, Kerr K, Kwiatkowski DJ, Ladanyi M, Nowak JA, Sholl L, Temple-Smolkin R, Solomon B, Souter LH, Thunnissen E, Tsao MS, Ventura CB, Wynes MW, Yatabe Y. Updated Molecular Testing Guideline for the Selection of Lung Cancer Patients for Treatment With Targeted Tyrosine Kinase Inhibitors: Guideline From the College of American Pathologists, the International Association for the Study of Lung Cancer, and the Association for Molecular Pathology. J Thorac Oncol. 2018 Mar;13(3):323-358. doi: 10.1016/j.jtho.2017.12.001. Epub 2018 Jan 25. PMID 29396253
- [Background] Faivre-Finn C, Vicente D, Kurata T, Planchard D, Paz-Ares L, Vansteenkiste JF, Spigel DR, Garassino MC, Reck M, Senan S, Naidoo J, Rimner A, Wu YL, Gray JE, Ozguroglu M, Lee KH, Cho BC, Kato T, de Wit M, Newton M, Wang L, Thiyagarajah P, Antonia SJ. Four-Year Survival With Durvalumab After Chemoradiotherapy in Stage III NSCLC-an Update From the PACIFIC Trial. J Thorac Oncol. 2021 May;16(5):860-867. doi: 10.1016/j.jtho.2020.12.015. Epub 2021 Jan 19. PMID 33476803
- [Background] Aredo JV, Mambetsariev I, Hellyer JA, Amini A, Neal JW, Padda SK, McCoach CE, Riess JW, Cabebe EC, Naidoo J, Abuali T, Salgia R, Loo BW Jr, Diehn M, Han SS, Wakelee HA. Durvalumab for Stage III EGFR-Mutated NSCLC After Definitive Chemoradiotherapy. J Thorac Oncol. 2021 Jun;16(6):1030-1041. doi: 10.1016/j.jtho.2021.01.1628. Epub 2021 Feb 12. PMID 33588109
- [Background] Guibert N, Pradines A, Favre G, Mazieres J. Current and future applications of liquid biopsy in nonsmall cell lung cancer from early to advanced stages. Eur Respir Rev. 2020 Feb 12;29(155):190052. doi: 10.1183/16000617.0052-2019. Print 2020 Mar 31. PMID 32051167
- [Background] Rolfo C, Mack PC, Scagliotti GV, Baas P, Barlesi F, Bivona TG, Herbst RS, Mok TS, Peled N, Pirker R, Raez LE, Reck M, Riess JW, Sequist LV, Shepherd FA, Sholl LM, Tan DSW, Wakelee HA, Wistuba II, Wynes MW, Carbone DP, Hirsch FR, Gandara DR. Liquid Biopsy for Advanced Non-Small Cell Lung Cancer (NSCLC): A Statement Paper from the IASLC. J Thorac Oncol. 2018 Sep;13(9):1248-1268. doi: 10.1016/j.jtho.2018.05.030. Epub 2018 Jun 6. PMID 29885479
- [Background] Heitzer E, Haque IS, Roberts CES, Speicher MR. Current and future perspectives of liquid biopsies in genomics-driven oncology. Nat Rev Genet. 2019 Feb;20(2):71-88. doi: 10.1038/s41576-018-0071-5. PMID 30410101
- [Background] Moding EJ, Liu Y, Nabet BY, Chabon JJ, Chaudhuri AA, Hui AB, Bonilla RF, Ko RB, Yoo CH, Gojenola L, Jones CD, He J, Qiao Y, Xu T, Heymach JV, Tsao A, Liao Z, Gomez DR, Das M, Padda SK, Ramchandran KJ, Neal JW, Wakelee HA, Loo BW Jr, Lin SH, Alizadeh AA, Diehn M. Circulating Tumor DNA Dynamics Predict Benefit from Consolidation Immunotherapy in Locally Advanced Non-Small Cell Lung Cancer. Nat Cancer. 2020 Feb;1(2):176-183. doi: 10.1038/s43018-019-0011-0. Epub 2020 Jan 20. PMID 34505064
- [Background] Dasari A, Morris VK, Allegra CJ, Atreya C, Benson AB 3rd, Boland P, Chung K, Copur MS, Corcoran RB, Deming DA, Dwyer A, Diehn M, Eng C, George TJ, Gollub MJ, Goodwin RA, Hamilton SR, Hechtman JF, Hochster H, Hong TS, Innocenti F, Iqbal A, Jacobs SA, Kennecke HF, Lee JJ, Lieu CH, Lenz HJ, Lindwasser OW, Montagut C, Odisio B, Ou FS, Porter L, Raghav K, Schrag D, Scott AJ, Shi Q, Strickler JH, Venook A, Yaeger R, Yothers G, You YN, Zell JA, Kopetz S. ctDNA applications and integration in colorectal cancer: an NCI Colon and Rectal-Anal Task Forces whitepaper. Nat Rev Clin Oncol. 2020 Dec;17(12):757-770. doi: 10.1038/s41571-020-0392-0. Epub 2020 Jul 6. PMID 32632268
- [Background] Pellini B, Chaudhuri AA. Circulating Tumor DNA Minimal Residual Disease Detection of Non-Small-Cell Lung Cancer Treated With Curative Intent. J Clin Oncol. 2022 Feb 20;40(6):567-575. doi: 10.1200/JCO.21.01929. Epub 2022 Jan 5. PMID 34985936
- [Background] Gale D, Heider K, Ruiz-Valdepenas A, Hackinger S, Perry M, Marsico G, Rundell V, Wulff J, Sharma G, Knock H, Castedo J, Cooper W, Zhao H, Smith CG, Garg S, Anand S, Howarth K, Gilligan D, Harden SV, Rassl DM, Rintoul RC, Rosenfeld N. Residual ctDNA after treatment predicts early relapse in patients with early-stage non-small cell lung cancer. Ann Oncol. 2022 May;33(5):500-510. doi: 10.1016/j.annonc.2022.02.007. Epub 2022 Mar 17. PMID 35306155
- [Background] Croitoru VM, Cazacu IM, Popescu I, Paul D, Dima SO, Croitoru AE, Tanase AD. Clonal Hematopoiesis and Liquid Biopsy in Gastrointestinal Cancers. Front Med (Lausanne). 2022 Jan 21;8:772166. doi: 10.3389/fmed.2021.772166. eCollection 2021. PMID 35127745
- [Background] Parikh AR, Van Seventer EE, Siravegna G, Hartwig AV, Jaimovich A, He Y, Kanter K, Fish MG, Fosbenner KD, Miao B, Phillips S, Carmichael JH, Sharma N, Jarnagin J, Baiev I, Shah YS, Fetter IJ, Shahzade HA, Allen JN, Blaszkowsky LS, Clark JW, Dubois JS, Franses JW, Giantonio BJ, Goyal L, Klempner SJ, Nipp RD, Roeland EJ, Ryan DP, Weekes CD, Wo JY, Hong TS, Bordeianou L, Ferrone CR, Qadan M, Kunitake H, Berger D, Ricciardi R, Cusack JC, Raymond VM, Talasaz A, Boland GM, Corcoran RB. Minimal Residual Disease Detection using a Plasma-only Circulating Tumor DNA Assay in Patients with Colorectal Cancer. Clin Cancer Res. 2021 Oct 15;27(20):5586-5594. doi: 10.1158/1078-0432.CCR-21-0410. Epub 2021 Apr 29. PMID 33926918